CLINICAL TRIAL: NCT03784092
Title: The Effect of Enhanced Mobility, Controlled Via Electronic Pedometers, During Induction of Labor by Extra Amniotic Balloon on Time to Delivery. A Randomized Controlled Trial
Brief Title: Effect Mobility During Induction of Labor on Time to Delivery. A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Noa Gonen, principal investigator, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0201-18-womc
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Labor Onset and Length Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention)
- feedback (Experimental)
  Interventions: Other: feedback

INTERVENTIONS:
Other: feedback — feedback by electronic pedometers regarding patient mobility while undergoing labor induction
  Arms: feedback

SUMMARY:
this is a andomized controlled trial the evaluates the effect of enhanced mobility, controlled via electronic pedometers, during induction of labor by extra amniotic balloon on time to delivery.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* low risk pregnancies
* singlelton
* vertex position
* undergoing labor induction with extra amniotic catheter
* no contraindication for enhanced mobility

Exclusion Criteria:

* medical recommendation for limited mobility
* status post cesarean delivery
* twin pregnancy
* premature rupture of membranes
* severe preeclampsia
* maternal comorbidity

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 224 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
time to delivery | labor ( catheter placement till delivery completion)
  time from extra amniotic catheter placement till delivery

IPD SHARING:
Plan to Share IPD: No